CLINICAL TRIAL: NCT01847261
Title: A Randomized, Controlled Double Blind Acute Study: Effects of Protein Blends on Muscle Protein Synthesis and Breakdown in Healthy Older Adults
Brief Title: Effects of Protein Blends on Muscle Protein Synthesis in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB #12-226
Record Dates: First submitted 2013-04-24; First posted 2013-05-06 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Muscle Synthesis
Keywords: soy; whey; muscle; older; mTOR; sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy Dairy Protein Blend (Experimental): 30 grams of Soy Dairy Protein Blend given as a single beverage following leg resistance exercise
  Interventions: Dietary Supplement: Soy Dairy Protein Blend
- Positive Control (Dairy Whey Protein) (Active Comparator): 30 grams of Dairy Whey Protein will be given as a single beverage following leg resistance exercise
  Interventions: Dietary Supplement: Positive Control (Dairy Whey Protein)

INTERVENTIONS:
Dietary Supplement: Soy Dairy Protein Blend
  Arms: Soy Dairy Protein Blend
Dietary Supplement: Positive Control (Dairy Whey Protein)
  Arms: Positive Control (Dairy Whey Protein)

SUMMARY:
During aging there is a tendency for muscle protein synthesis (growth) to become less efficient and the resulting consequence leads to reduced muscle mass (sarcopenia) which can affect strength and mobility. Protein consumption may be one opportunity to alleviate this problem especially when consumed in appropriate amounts following resistance training. This study is designed to determine if a soy dairy protein blend, shown to be effective in younger adults, will produce beneficial muscle protein synthesis in older healthy adults following resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

55-70 yr olds Stable Body weight

Exclusion Criteria:

1. Exercise training (>2 weekly sessions of moderate to high intensity aerobic or resistance exercise)
2. Significant heart, liver, kidney, blood, respiratory disease or thyroid issues
3. Peripheral vascular disease
4. Orthopedic injury that prohibits participation in the exercise training
5. Diabetes mellitus or other untreated endocrine disease
6. Active cancer (all groups) and history of cancer
7. Acute infectious disease or history of chronic infections (e.g. TB, hepatitis, HIV, herpes)
8. Neurologic Injury or disease
9. Recent (within 6 months) treatment with anabolic steroids, or corticosteroids.
10. Alcohol or drug abuse
11. Tobacco use (smoking or chewing)
12. Malnutrition (BMI < 20 kg/m2, hypoalbuminemia, and/or hypotransferrinemia)
13. Obesity (BMI > 30 kg/m2)
14. Low hemoglobin levels (below normal values)
15. Food allergies
16. Taking dietary supplements such as green tea, omega 3 fatty acids, etc.
17. Females

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fractional Synthetic Rate (Muscle Protein Synthesis) | baseline, 3 hrs, 5 hrs
  The fractional synthesis rate (FSR) of mixed muscle proteins will be calculated from the incorporation rate of L-[ring-13C6]Phenylalanine into the mixed muscle proteins, and the free-tissue phenylalanine enrichment.

SECONDARY OUTCOMES:
Anti-inflammatory and Anti-oxidant Markers | baseline, 3 hrs, 5 hrs
  Proteins will be assessed that are markers of oxidative damage and inflammation (NFkB, IL-1, IL-6) and proteolysis (MuRF, MAFBx).
Intracellular Signalling Genes and Proteins | baseline, 3 hrs, 5 hrs
  Phosphorylation of Mammalian Target of Rapamycin (mTOR) pathway will be measured using Western blot techniques

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Borack MS, Reidy PT, Husaini SH, Markofski MM, Deer RR, Richison AB, Lambert BS, Cope MB, Mukherjea R, Jennings K, Volpi E, Rasmussen BB. Soy-Dairy Protein Blend or Whey Protein Isolate Ingestion Induces Similar Postexercise Muscle Mechanistic Target of Rapamycin Complex 1 Signaling and Protein Synthesis Responses in Older Men. J Nutr. 2016 Dec;146(12):2468-2475. doi: 10.3945/jn.116.231159. Epub 2016 Oct 26. PMID 27798330